CLINICAL TRIAL: NCT02780193
Title: Open Protocol for the Use of an Intravenous Fat Emulsion Comprised of Fish Oils (Omegaven) in the Treatment of Parenteral Nutrition (PN) Induced Liver Injury
Brief Title: Intravenous Fish Oils in the Treatment of Parenteral Nutrition Liver Injury
Status: Approved for marketing | Type: Expanded Access
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Aloka Patel, Associate Professor, Rush University Medical Center
Other Study IDs: 14051906
Record Dates: First submitted 2015-05-22; First posted 2016-05-23 (Estimated); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Cholestasis; Total Parenteral Nutrition-induced Cholestasis
MeSH Terms: conditions — Cholestasis | interventions — fish oil triglycerides

INTERVENTIONS:
Drug: Omegaven — Therapy with Omegaven® will be initiated and maintained at 1 g/kg/day. It will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition. If additional non-protein calories are needed, they will be provided as carbohydrates. No other parenteral form of fat emulsion will be used during Omegaven® therapy.The Omegaven® dose may be discontinued if the subject is receiving adequate enteral nutrition to meet metabolic and growth needs.

SUMMARY:
The purpose of this study is to provide intravenous omega-3 fatty acids and monitor tolerance in subjects with prolonged parenteral nutrition dependence and parenteral nutrition-associated cholestasis through expanded access.

DETAILED DESCRIPTION:
Therapy with Omegaven will be initiated and maintained at 1 g/kg/day in subjects with parenteral nutrition-associated cholestasis and prolonged parenteral nutrition dependence who qualify for expanded access. It will be infused intravenously through either a central or peripheral catheter in conjunction with parenteral nutrition. If additional non-protein calories are needed, they will be provided as carbohydrates. No other parenteral form of fat emulsion will be used during Omegaven therapy unless the subject is not receiving adequate calories and additional dextrose may not be administered to the subject because of severe persistent hyperglycemia, respiratory compromise, or other clinical conditions, or unless the patient develops essential fatty acid deficiency as confirmed by laboratory parameters. The same standards of care provided to all subjects receiving parenteral nutrition solution will be followed.

Regular PN monitoring will be accomplished by analyzing clinical and laboratory parameters, including serum electrolytes, hematological studies, renal function, hepatic function, blood clotting factors, protein and nutrition status and trace mineral status. An essential fatty acid profile and lipid panel will be sampled from the subject to monitor the effects of Omegaven.

Blood will be sampled for an essential fatty acid profile and lipid panel before beginning Omegaven, weekly while the patient is on Omegaven and has a direct (conjugated) bilirubin ≥ 2 mg/dL, and then monthly while the patient is on Omegaven and has a direct (conjugated) bilirubin < 2 mg/dL. Subjects will also be monitored daily for clinical signs and symptoms of essential fatty acid deficiency, including dermatitis and hair loss.

Dose reduction and titration or discontinuation will occur if there is evidence of hypertriglyceridemia (serum triglycerides > 200 mg/dL), allergic response, toxicity or evidence of bleeding that is believed to be caused or worsened by Omegaven. If lipid intolerance develops, defined as serum triglyceride level > 200 mg/dL, lipids will be stopped for at least 4 hours and a repeat serum triglyceride level will be obtained. If the triglycerides continue to remain high a dosage reduction of 25% of the current dose will be considered. Growth indices include weight, length, and head circumference will also be monitored. The Omegaven dose may be discontinued if the subject is receiving adequate enteral nutrition to meet metabolic and growth needs.

Subjects will receive follow-up visits per the customary medical (GI) or surgical follow-up schedule for a period of 36 months after discontinuation of Omegaven. Follow up visits will occur at least annually, but may be more frequent based on the subjects' tolerance of and weight gain on enteral nutrition.

As previously mentioned, Omegaven will be infused in the same manner as conventional fat emulsions through either a central or peripheral line. The emulsion is isotonic. It is compatible with parenteral nutrition solutions and may be co-infused via y-site. Source containers will be changed every 24 hours and unused product discarded. Omegaven may be infused through a 1.2 micron inline filter.

ELIGIBILITY:
Inclusion Criteria:

Patients from birth to 18 years of age who:

* are receiving PN,
* are predicted to receive at least another 30 days of PN, and
* have liver disease with at least a serum direct (conjugated) bilirubin ≥ 2 mg/dL

  * Patients from birth to 18 years of age who have a soybean allergy (per parental report) and require parenteral fat
  * Patients with significant liver disease due to parenteral nutrition despite utilization of all appropriate conventional therapies.
  * Signed patient/parent informed consent
  * Hospitalized due to medical or surgical condition prior to Omegaven initiation

Exclusion Criteria:

* Those who do not fulfill the inclusion criteria
* Those who choose not to consent to the study
* Those in whom 3rd party funding is not secured to support this investigational treatment
* Known fish or egg protein allergy (per parental report)
* All other causes of liver disease (cystic fibrosis, biliary atresia, and alpha 1 anti- trypsin deficiency)
* Severe hemorrhagic disorders (platelet count below 50000)
* Collapse and shock
* Embolism
* Undefined coma status
* Impaired lipid metabolism (serum triglycerides > 200 mg/dL on 1 g/kg/day intralipid)
* Unstable diabetes mellitus
* Stroke
* Recent cardiac infarction

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Aloka L Patel, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Puder M, Valim C, Meisel JA, Le HD, de Meijer VE, Robinson EM, Zhou J, Duggan C, Gura KM. Parenteral fish oil improves outcomes in patients with parenteral nutrition-associated liver injury. Ann Surg. 2009 Sep;250(3):395-402. doi: 10.1097/SLA.0b013e3181b36657. PMID 19661785
- [Background] Gura KM, Lee S, Valim C, Zhou J, Kim S, Modi BP, Arsenault DA, Strijbosch RA, Lopes S, Duggan C, Puder M. Safety and efficacy of a fish-oil-based fat emulsion in the treatment of parenteral nutrition-associated liver disease. Pediatrics. 2008 Mar;121(3):e678-86. doi: 10.1542/peds.2007-2248. PMID 18310188